CLINICAL TRIAL: NCT05283057
Title: Effect of Sodium Glucose Transporter 2 Inhibitor Empagliflozin on Proteinuria and Kidney Disease Progression in Patients With Non-diabetic Glomerulonephritis- A Randomized Controlled Trial
Brief Title: Empagliflozin in Patients With Glomerulonephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA-21-297
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Glomerulonephritis; Proteinuria
Keywords: sodium glucose cotransporter inhibitors; Empagliflozin
MeSH Terms: conditions — Glomerulonephritis; Proteinuria | interventions — empagliflozin; 5'-palmitoyl cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Empagliflozin (Active Comparator): 25 patients with glomerulonephritis and proteinuria who were treated with Empagliflozin
  Interventions: Drug: Empagliflozin 25 MG
- Group 2: (Placebo Comparator): 25 patients with glomerulonephritis and proteinuria who were treated with standard treatment and placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — single dose of the SGLT inhibitor Empagliflozin was given
  Other Names: EMPA
  Arms: Group 1: Empagliflozin
Drug: placebo — single dose of placebo that is similar to Empagliflozin in physical appearance
  Other Names: PLAC
  Arms: Group 2:

SUMMARY:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors are newly developed antihyperglycemic medications. In addition to their glucose lowering properties, they have been shown to have favourable effects on the cardiovascular and renal outcome in patients with diabetes. one of the most interesting renal effects is reduction of proteinuria. The aim of our study was examine the effect of SGLT inhibitors on proteinuria in patients with glomerulonephritis. This study is a randomised controlled trial.

DETAILED DESCRIPTION:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors are newly developed antihyperglycemic medications. In addition to their glucose lowering properties, they have been shown to have favourable effects on the cardiovascular and renal outcome in patients with diabetes.The favourable cardiovascular effects include increased diuresis , reduction of blood pressure and reduction of hospitalisation for heart failure one of the most interesting renal effects is reduction of proteinuria. The aim of our study was examine the effect of SGLT inhibitors on proteinuria in patients with glomerulonephritis. This study is a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years.
2. Urinary protein excretion > 500 mg/g and eGFR ≥ 30 mL/min/1.73 m2 (CKD stages 1-3).
3. On a stable dose of an ACEi or ARBs together with their immunosuppression protocol for at least 4 weeks prior to randomization.
4. Who signed informed consent.
5. Women of Child-Bearing Potential (WOCBP) used an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug in such a manner that the risk of pregnancy was minimized.

Exclusion Criteria:

* a) Diagnosis of type 1 or type 2 diabetes mellitus b) Urinary protein excretion of less than 500 mg/g and eGFR < 30 ml/min

  * 1.7m2 c) Active malignancy d) Any medication, surgical or medical condition that may significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following: History of active inflammatory bowel disease within the last six months; Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last six months; Pancreatic injury or pancreatitis within the last six months.

    e) Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3x ULN at the screening visit, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt.

    f) Evidence of urinary tract obstruction. g) History of hypersensitivity or contraindications to empagliflozin. h) Subject who, in the assessment of the investigator, may be at risk for dehydration or volume depletion that may affect the interpretation of efficacy or safety data.

    i) Participation in any clinical investigation within 3 months prior to initial dosing.

    j) History of noncompliance to medical regimens or unwillingness to comply with the study protocol.

    k) Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
protein to creatinine ratio | 3 months
  measurement of urinary protein to creatinine ratio as a marker of proteinuria

SECONDARY OUTCOMES:
Decline of glomerular filtration rate | 3 months
  Decline in estimated glomerular filtration rate over

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelaziz, PHD, Principal Investigator — Kasr Alainy faculty of medicine
Locations (1):
- Cairo university hospitals, Cairo, Egypt